CLINICAL TRIAL: NCT01122290
Title: Inducing Preschool Children's Emotional Eating: Relationships With Parental Feeding Practices.
Brief Title: Inducing Children's Emotional Eating
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: Loughborough University (Other)
Responsible Party: Dr Jackie Blissett, School of Psychology, University of Birmingham
Other Study IDs: H10543 (Lboro)
Record Dates: First submitted 2010-05-12; First posted 2010-05-13 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Emotional Eating Behaviour
Keywords: Emotional eating; Eating in the absence of hunger; emotion induction
MeSH Terms: conditions — Emotional Eating

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- negative emotion: Children experienced induction of mild negative emotion through a jigsaw with a missing piece (negative emotion group)
- neutral emotion: Vs. Same task with No missing piece (neutral emotion).

SUMMARY:
Background: Children's emotional eating is related to greater BMI and less healthy diet but little is known about the early development of this behavior.

Objective: This study aimed to examine the relationships between preschool children's emotional eating and parental feeding practices using experimental manipulation of child mood and food intake in a laboratory setting.

Design: 25 3-5 year old children and their mothers sat together and ate a standard meal to satiety. Mothers completed questionnaires about their feeding practices. Children were assigned to a control or negative mood condition. Children's consumption of snack foods in the absence of hunger was measured.

ELIGIBILITY:
Inclusion Criteria:

* Child age between 3 years and 5 years
* No disease/disorder affecting eating
* No learning disability

Exclusion Criteria:

* Any child brought in by a (non-primary care-giving) grandparent
* Child BMI at extreme of sample
* Incongruous mood shift to condition
* Child of non-english speaking/reading parent

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy 3-5 year old children in the UK (within approx. radius of 10 miles of Loughborough University).
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
eating in the absence of hunger | @ 60 minutes into study, at ~4 years of age
  Child's consumption of kcal from snack foods in the absence of hunger

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sport, Exercise and Health Sciences, Loughborough University, Loughborough, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Farrow CV, Haycraft E, Blissett JM. Teaching our children when to eat: how parental feeding practices inform the development of emotional eating--a longitudinal experimental design. Am J Clin Nutr. 2015 May;101(5):908-13. doi: 10.3945/ajcn.114.103713. Epub 2015 Mar 18. PMID 25787999
- [Derived] Blissett J, Haycraft E, Farrow C. Inducing preschool children's emotional eating: relations with parental feeding practices. Am J Clin Nutr. 2010 Aug;92(2):359-65. doi: 10.3945/ajcn.2010.29375. Epub 2010 Jun 9. PMID 20534744